CLINICAL TRIAL: NCT01183013
Title: A Randomised, Double-blind Parallel Group Study to Compare the Efficacy and Safety of Initial Combination Therapy With Linagliptin 5 mg + Pioglitazone 15 mg, 30 mg, or 45 mg, vs. Monotherapy With Pioglitazone (15 mg, 30 mg, or 45 mg) or Linagliptin 5 mg Once Daily for 30 Weeks, Followed by a Blinded Trial Period on Linagliptin 5 mg + Pioglitazone 30 or 45 mg Versus Pioglitazone Monotherapy 30 or 45 mg or Linagliptin 5 mg for up to 54 Weeks in Type 2 Diabetic Patients With Insufficient Glycaemic Control on Diet and Exercise
Brief Title: 30 Week Parallel Group Comparison Study of Linagliptin + Pioglitazone (5+15, 5+30 and 5+45 mg) qd Versus Respective Monotherapies, Followed by a Comparison of 5mg+30mg and 5mg+45mg Versus Respective Monotherapies in Type 2 Diabetes for up to 54 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1264.3; 2008-008127-15 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Linagliptin

ARMS (7):
- Pioglitazone 15 mg (Active Comparator): Pioglitazone Capsules 15 mg once daily
  Interventions: Drug: Pioglitazone 15 mg
- Pioglitazone 30 mg (Active Comparator): Pioglitazone Capsules 30 mg once daily
  Interventions: Drug: Pioglitazone 30 mg
- Pioglitazone 45 mg (Active Comparator): Pioglitazone Capsules 45 mg once daily
  Interventions: Drug: Pioglitazone 45 mg
- Linagliptin 5mg (Active Comparator): Linagliptin 5mg Tablets once daily
  Interventions: Drug: Linagliptin 5mg
- Linagliptin 5mg / Pioglitazone 15 mg (Experimental): Linagliptin 5mg / Pioglitazone 15 mg Tablets once daily
  Interventions: Drug: Linagliptin 5mg / Pioglitazone 15 mg FDC
- Linagliptin 5mg / Pioglitazone 30 mg (Experimental): Linagliptin 5mg / Pioglitazone 30 mg Tablets once daily
  Interventions: Drug: Linagliptin 5mg / Pioglitazone 30 mg FDC
- Linagliptin 5mg / Pioglitazone 45 mg (Experimental): Linagliptin 5mg / Pioglitazone 45 mg Tablets once daily
  Interventions: Drug: Linagliptin 5mg / Pioglitazone 45 mg FDC

INTERVENTIONS:
Drug: Pioglitazone 15 mg — Pioglitazone Capsules 15 mg once daily for 30 weeks followed by Pioglitazone Capsules 30 mg once daily for up to 54 weeks
  Arms: Pioglitazone 15 mg
Drug: Pioglitazone 45 mg — Pioglitazone Capsules 30 mg once daily for 6 weeks followed by Pioglitazone Capsules 45 mg once daily for up to 78 weeks
  Arms: Pioglitazone 45 mg
Drug: Pioglitazone 30 mg — Pioglitazone Capsules 30 mg once daily for up to 84 weeks
  Arms: Pioglitazone 30 mg
Drug: Linagliptin 5mg / Pioglitazone 45 mg FDC — Linagliptin 5mg low dose / Pioglitazone 30 mg Tablets once daily for 6 weeks followed by Linagliptin 5mg low dose / Pioglitazone 45 mg FDC Tablets once daily for up to 78 weeks
  Arms: Linagliptin 5mg / Pioglitazone 45 mg
Drug: Linagliptin 5mg / Pioglitazone 30 mg FDC — Linagliptin 5mg low dose / Pioglitazone 30 mg FDC Tablets once daily for up to 84 weeks
  Arms: Linagliptin 5mg / Pioglitazone 30 mg
Drug: Linagliptin 5mg — Linagliptin 5mg Tablets low dose once daily for 30 weeks followed by Linagliptin 5mg low dose / Pioglitazone 30 mg FDC Tablets once daily for up to 54 weeks
  Arms: Linagliptin 5mg
Drug: Linagliptin 5mg / Pioglitazone 15 mg FDC — Linagliptin 5mg low dose / Pioglitazone 15 mg FDC Tablets once daily for 30 weeks followed by Linagliptin 5mg low dose / Pioglitazone 30 mg FDC Tablets once daily for up to 54 weeks
  Arms: Linagliptin 5mg / Pioglitazone 15 mg

SUMMARY:
The primary objective is to demonstrate superior glycaemic control (HbA1c reduction) after 30 weeks of linagliptin/pioglitazone (5/15, 5/30 and 5/45 mg) versus the respective individual monotherapies of pioglitazone (15 mg, 30 mg, or 45 mg, administered orally once daily), and linagliptin (5 mg, administered orally once daily). In addition, durability of treatment effect and safety under chronic treatment conditions will be investigated.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus prior to informed consent
2. Male and female patients with insufficient glycaemic control (HbA1c >= 7.0 to <= 10.5% at Visit 2) on diet and exercise alone, without oral antidiabetic drug therapy within 10 weeks prior to start of the run-in period (date of Visit 2)
3. Age >= 18 and <= 80 years at start date of Visit 1 (Screening)
4. BMI <= 45 kg/m2 (Body Mass Index) at start date of Visit 1 (Screening)
5. Signed and dated written informed consent by start date of Visit 1 in accordance with GCP and local legislation

Exclusion criteria:

1. Uncontrolled hyperglycaemia with a confirmed glucose level > 240 mg/dl (> 13.3 mmol/l) after an overnight fast during screening or placebo run-in period (cf. Section 3.3.4.1)
2. Myocardial infarction within 6 months, stroke or TIA within 3 months prior to informed consent
3. Clinical evidence of active liver disease (e.g. jaundice) or the ALT level > 2.5 times the upper limit of normal (according to pioglitazone label)
4. Bariatric surgery, performed within the past 2 years prior to informed consent or planned at the time of informed consent
5. Gastrointestinal surgeries prior to informed consent that induce chronic malabsorption
6. Known hypersensitivity or allergy to the investigational products (linagliptin and/or pioglitazone) or their excipients (including matching placebos)
7. Contraindications to pioglitazone as defined in the local prescribing information (SPC), particularly :

   * Diagnose of heart failure or history of heart failure
   * Haemodialysis patients, due to limited experience with pioglitazone
8. Treatment with gemfibrozil, montelukast, trimethoprim, or rifampicin - according to pioglitazone label and respective restrictions in Section 4.2.2
9. Treatment with rosiglitazone, pioglitazone, GLP-1 analogues, or insulin within 3 months prior to informed consent
10. Treatment with anti-obesity drugs (e.g. sibutramine, orlistat) 3 months prior to informed consent
11. Alcohol or drug abuse within the 3 months prior to informed consent or history of alcoholism
12. Current treatment with systemic corticosteroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent
13. Participation in another trial with an investigational drug within 30 days prior to informed consent
14. Any other clinical condition as judged by the investigator that would not allow the safe completion of the protocol, e.g. inability of patients to comply with study procedures
15. Pre-menopausal women (last menstruation <= 1 year prior to informed consent) who:

    * are nursing or pregnant or
    * are of child-bearing potential (i.e. not permanently sterilised) and are not practicing a highly effective method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial.

    A highly effective method of birth control is defined - according to the Note for Guidance on non-clinical safety studies for the conduct of human trials for pharmaceuticals (CPMP/ICH/286/95, modification) - as those which result in a low failure rate (i. e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal intrauterine devices/systems (IUDs/IUSs), sexual abstinence or vasectomised partner
16. Symptomatic gallbladder disease in the last six months
17. Medical history of pancreatitis.
18. Patients with urinary bladder cancer or a history of urinary bladder cancer or uninvestigated macroscopic haematuria
19. Any other contraindication or restriction for use of pioglitazone in accordance with the local prescribing information for pioglitazone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Actual)
Dates: Start 2010-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (132):
- United States (74):
  - 1264.3.01026 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1264.3.01021 Boehringer Ingelheim Investigational Site, Montgomery, Alabama
  - 1264.3.01020 Boehringer Ingelheim Investigational Site, Muscle Shoals, Alabama
  - 1264.3.01062 Boehringer Ingelheim Investigational Site, Chandler, Arizona
  - 1264.3.01064 Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - 1264.3.01049 Boehringer Ingelheim Investigational Site, Carmichael, California
  - 1264.3.01078 Boehringer Ingelheim Investigational Site, Chino, California
  - 1264.3.01031 Boehringer Ingelheim Investigational Site, Concord, California
  - 1264.3.01037 Boehringer Ingelheim Investigational Site, Lakewood, California
  - 1264.3.01065 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1264.3.01006 Boehringer Ingelheim Investigational Site, Norwalk, California
  - 1264.3.01001 Boehringer Ingelheim Investigational Site, Rancho Cucamonga, California
  - 1264.3.01059 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1264.3.01023 Boehringer Ingelheim Investigational Site, Tarzana, California
  - 1264.3.01016 Boehringer Ingelheim Investigational Site, Tustin, California
  - 1264.3.01058 Boehringer Ingelheim Investigational Site, Valencia, California
  - 1264.3.01083 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 1264.3.01027 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1264.3.01033 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 1264.3.01035 Boehringer Ingelheim Investigational Site, Boca Raton, Florida
  - 1264.3.01015 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1264.3.01082 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1264.3.01036 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1264.3.01013 Boehringer Ingelheim Investigational Site, Longwood, Florida
  - 1264.3.01038 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1264.3.01042 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1264.3.01079 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1264.3.01019 Boehringer Ingelheim Investigational Site, Port Orange, Florida
  - 1264.3.01018 Boehringer Ingelheim Investigational Site, Saint Cloud, Florida
  - 1264.3.01009 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1264.3.01012 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1264.3.01008 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1264.3.01055 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1264.3.01061 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1264.3.01074 Boehringer Ingelheim Investigational Site, Blue Ridge, Georgia
  - 1264.3.01084 Boehringer Ingelheim Investigational Site, Cartersville, Georgia
  - 1264.3.01060 Boehringer Ingelheim Investigational Site, Perry, Georgia
  - 1264.3.01050 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 1264.3.01077 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1264.3.01052 Boehringer Ingelheim Investigational Site, Brownsburg, Indiana
  - 1264.3.01075 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1264.3.01076 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1264.3.01073 Boehringer Ingelheim Investigational Site, Franklin, Indiana
  - 1264.3.01002 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1264.3.01007 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1264.3.01010 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 1264.3.01028 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1264.3.01029 Boehringer Ingelheim Investigational Site, Sunset, Louisiana
  - 1264.3.01069 Boehringer Ingelheim Investigational Site, Hyattsville, Maryland
  - 1264.3.01066 Boehringer Ingelheim Investigational Site, Southfield, Michigan
  - 1264.3.01057 Boehringer Ingelheim Investigational Site, Great Falls, Montana
  - 1264.3.01045 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 1264.3.01044 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1264.3.01022 Boehringer Ingelheim Investigational Site, Zanesville, Ohio
  - 1264.3.01032 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1264.3.01051 Boehringer Ingelheim Investigational Site, Fleetwood, Pennsylvania
  - 1264.3.01025 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1264.3.01081 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1264.3.01003 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1264.3.01011 Boehringer Ingelheim Investigational Site, Kingsport, Tennessee
  - 1264.3.01017 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 1264.3.01067 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1264.3.01004 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1264.3.01039 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1264.3.01041 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1264.3.01047 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1264.3.01070 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1264.3.01040 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1264.3.01048 Boehringer Ingelheim Investigational Site, Midland, Texas
  - 1264.3.01030 Boehringer Ingelheim Investigational Site, New Braunfels, Texas
  - 1264.3.01071 Boehringer Ingelheim Investigational Site, North Richland Hills, Texas
  - 1264.3.01085 Boehringer Ingelheim Investigational Site, Plano, Texas
  - 1264.3.01046 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1264.3.01056 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
- Estonia (10):
  - 1264.3.37207 Boehringer Ingelheim Investigational Site, Harju
  - 1264.3.37209 Boehringer Ingelheim Investigational Site, Pärnu
  - 1264.3.37201 Boehringer Ingelheim Investigational Site, Tallinn
  - 1264.3.37202 Boehringer Ingelheim Investigational Site, Tallinn
  - 1264.3.37203 Boehringer Ingelheim Investigational Site, Tallinn
  - 1264.3.37204 Boehringer Ingelheim Investigational Site, Tallinn
  - 1264.3.37205 Boehringer Ingelheim Investigational Site, Tallinn
  - 1264.3.37208 Boehringer Ingelheim Investigational Site, Tallinn
  - 1264.3.37206 Boehringer Ingelheim Investigational Site, Tartu
  - 1264.3.37210 Boehringer Ingelheim Investigational Site, Viljandi County
- Germany (10):
  - 1264.3.49001 Boehringer Ingelheim Investigational Site, Bad Lauterberg / Harz
  - 1264.3.49007 Boehringer Ingelheim Investigational Site, Dietzenbach
  - 1264.3.49002 Boehringer Ingelheim Investigational Site, Dortmund
  - 1264.3.49009 Boehringer Ingelheim Investigational Site, Essen
  - 1264.3.49003 Boehringer Ingelheim Investigational Site, Hamburg
  - 1264.3.49012 Boehringer Ingelheim Investigational Site, Ingelheim
  - 1264.3.49008 Boehringer Ingelheim Investigational Site, Leipzig
  - 1264.3.49005 Boehringer Ingelheim Investigational Site, Mainz
  - 1264.3.49010 Boehringer Ingelheim Investigational Site, Offenbach
  - 1264.3.49004 Boehringer Ingelheim Investigational Site, Stuhr
- Latvia (13):
  - 1264.3.37105 Boehringer Ingelheim Investigational Site, Daugavpils
  - 1264.3.37112 Boehringer Ingelheim Investigational Site, Daugavpils
  - 1264.3.37113 Boehringer Ingelheim Investigational Site, Daugavpils
  - 1264.3.37110 Boehringer Ingelheim Investigational Site, Jelgava
  - 1264.3.37101 Boehringer Ingelheim Investigational Site, Liepāja
  - 1264.3.37106 Boehringer Ingelheim Investigational Site, Ogre
  - 1264.3.37104 Boehringer Ingelheim Investigational Site, Riga
  - 1264.3.37108 Boehringer Ingelheim Investigational Site, Riga
  - 1264.3.37109 Boehringer Ingelheim Investigational Site, Riga
  - 1264.3.37111 Boehringer Ingelheim Investigational Site, Riga
  - 1264.3.37107 Boehringer Ingelheim Investigational Site, Talsi
  - 1264.3.37102 Boehringer Ingelheim Investigational Site, Tukums
  - 1264.3.37103 Boehringer Ingelheim Investigational Site, Valmiera
- Spain (12):
  - 1264.3.34013 Boehringer Ingelheim Investigational Site, Badía Del Vallès - Barcelona
  - 1264.3.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1264.3.34008 Boehringer Ingelheim Investigational Site, Barcelona
  - 1264.3.34005 Boehringer Ingelheim Investigational Site, Borges Del Camp- Tarragona
  - 1264.3.34006 Boehringer Ingelheim Investigational Site, Canet de Mar - Barcelona
  - 1264.3.34010 Boehringer Ingelheim Investigational Site, Centelles - Barcelona
  - 1264.3.34009 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1264.3.34004 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat - Barcelona
  - 1264.3.34002 Boehringer Ingelheim Investigational Site, Sant Adrià Del Besós- Barcelona
  - 1264.3.34007 Boehringer Ingelheim Investigational Site, Tarrega - Lleida
  - 1264.3.34012 Boehringer Ingelheim Investigational Site, Valencia
  - 1264.3.34011 Boehringer Ingelheim Investigational Site, Vic - Barcelona
- United Kingdom (13):
  - 1264.3.44032 Boehringer Ingelheim Investigational Site, Annan
  - 1264.3.44028 Boehringer Ingelheim Investigational Site, Ash Vale, Aldershot
  - 1264.3.44029 Boehringer Ingelheim Investigational Site, Baillieston, Glasgow
  - 1264.3.44008 Boehringer Ingelheim Investigational Site, Balham
  - 1264.3.44021 Boehringer Ingelheim Investigational Site, Bradford-on-Avon
  - 1264.3.44019 Boehringer Ingelheim Investigational Site, Burbage
  - 1264.3.44012 Boehringer Ingelheim Investigational Site, Chesterfield
  - 1264.3.44027 Boehringer Ingelheim Investigational Site, Chestfield, Whitstable
  - 1264.3.44011 Boehringer Ingelheim Investigational Site, Chippenham
  - 1264.3.44033 Boehringer Ingelheim Investigational Site, Johnstone
  - 1264.3.44007 Boehringer Ingelheim Investigational Site, Midsomer Norton
  - 1264.3.44034 Boehringer Ingelheim Investigational Site, Paisley
  - 1264.3.44031 Boehringer Ingelheim Investigational Site, Warminster

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After Amendment #5, patients were considered COMPLETED at the end of Part A (30 weeks) or after their next Part B visit (up to 54 weeks) if already in Part B. Before Amendment #5, all patients were considered COMPLETED at the end of Part A + Part B (84 weeks).
Groups:
- Pio15/Pio30: Participants treated with pioglitazone 15mg for 30 weeks followed by pioglitazone 30mg for up to 54 weeks.
- Pio30/Pio30: Participants treated with pioglitazone 30mg for 30 weeks followed by pioglitazone 30mg for up to 54 weeks.
- Pio45/Pio45: Participants treated with pioglitazone 30 mg for 6 weeks and then were titrated up to pioglitazone 45mg for 24 weeks followed by pioglitazone 45mg for up to 54 weeks.
- Lina5/Lina5: Participants treated with linagliptin 5mg once daily for 30 weeks followed by linagliptin 5mg once daily for up to 54 weeks.
- Lina5Pio15/Lina5Pio30: Participants treated with linagliptin 5mg + pioglitazone 15mg fixed dose combination (FDC) for 30 weeks followed by linagliptin 5mg + pioglitazone 30mg FDC for up to 54 weeks.
- Lina5Pio30/Lina5Pio30: Participants treated with linagliptin 5mg + pioglitazone 30mg fixed dose combination (FDC) for 30 weeks followed by linagliptin 5mg + pioglitazone 30mg FDC for up to 54 weeks.
- Lina5Pio45/Lina5Pio45: Participants treated with linagliptin 5mg + pioglitazone 30mg fixed dose combination (FDC) for 6 weeks and linagliptin 5mg + pioglitazone 45mg FDC for 24 weeks followed by linagliptin 5mg + pioglitazone 45mg FDC for up to 54 weeks.
Period: Overall Study
Arm/Group | Pio15/Pio30 | Pio30/Pio30 | Pio45/Pio45 | Lina5/Lina5 | Lina5Pio15/Lina5Pio30 | Lina5Pio30/Lina5Pio30 | Lina5Pio45/Lina5Pio45
Started | 131 | 140 | 138 | 135 | 126 | 133 | 133
Completed | 86 (Completed is first 30 weeks (Part A) or up to 84 weeks in relation to Protocol Amendment #5) | 101 (Completed is first 30 weeks (Part A) or up to 84 weeks in relation to Protocol Amendment #5) | 97 (Completed is first 30 weeks (Part A) or up to 84 weeks in relation to Protocol Amendment #5) | 105 (Completed is first 30 weeks (Part A) or up to 84 weeks in relation to Protocol Amendment #5) | 90 (Completed is first 30 weeks (Part A) or up to 84 weeks in relation to Protocol Amendment #5) | 88 (Completed is first 30 weeks (Part A) or up to 84 weeks in relation to Protocol Amendment #5) | 96 (Completed is first 30 weeks (Part A) or up to 84 weeks in relation to Protocol Amendment #5)
Not Completed | 45 | 39 | 41 | 30 | 36 | 45 | 37
Not completed — Adverse Event | 6 | 8 | 5 | 5 | 10 | 10 | 6
Not completed — Lack of Efficacy | 3 | 2 | 1 | 2 | 1 | 2 | 0
Not completed — Protocol Violation | 5 | 2 | 4 | 0 | 4 | 3 | 3
Not completed — Lost to Follow-up | 7 | 3 | 4 | 3 | 2 | 6 | 5
Not completed — Withdrawal by Subject | 9 | 13 | 10 | 8 | 7 | 9 | 10
Not completed — Reasons other than stated above | 15 | 11 | 17 | 12 | 12 | 15 | 13

BASELINE CHARACTERISTICS:
Population: All patients from the Full Analysis Set (FAS) which includes those patients in the treated set who had a baseline HbA1c value and at least one on-treatment HbA1c value.
Groups:
- Lina5/Lina5: Participants treated with linagliptin 5mg + pioglitazone 15mg fixed dose combination (FDC) for 30 weeks followed by linagliptin 5mg + pioglitazone 30mg FDC for up to 54 weeks.
- Lina5Pio15/Lina5Pio30: Participants treated with linagliptin 5mg + pioglitazone 15mg fixed dose combination (FDC) for 30 weeks followed by a blinded trial period on linagliptin 5mg + pioglitazone 30mg FDC
- Total: Total of all reporting groups
Arm/Group | Pio15/Pio30 | Pio30/Pio30 | Pio45/Pio45 | Lina5/Lina5 | Lina5Pio15/Lina5Pio30 | Lina5Pio30/Lina5Pio30 | Lina5Pio45/Lina5Pio45 | Total
Number analyzed (Participants) | 124 | 134 | 134 | 130 | 120 | 125 | 126 | 893
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.4) | 57.2 (11.1) | 56.5 (11.1) | 56.3 (10.1) | 57.1 (10.2) | 56.4 (10.0) | 60.1 (10.2) | 57.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 64 | 66 | 51 | 54 | 61 | 57 | 410
  Male | 67 | 70 | 68 | 79 | 66 | 64 | 69 | 483
Baseline HbA1c [Mean (Standard Deviation); unit: percent] | 8.33 (0.93) | 7.99 (0.85) | 8.12 (0.87) | 8.01 (0.88) | 8.13 (0.94) | 8.17 (1.07) | 8.01 (0.81) | 8.11 (0.91)
Baseline fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 171.3 (39.3) | 165.8 (40.0) | 167.5 (37.9) | 161.4 (38.1) | 167.3 (39.5) | 168.8 (46.8) | 162.3 (36.8) | 166.3 (39.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c After 30 Weeks of Treatment.
Description: HbA1c is measured as a percentage. The change from baseline is the Week 30 HbA1c minus the baseline HbA1c.
Time Frame: Baseline and 30 weeks
Population: Patients from Full Analysis Set (FAS) with last observation carried forward (LOCF) used to handle missing values at Week 30. FAS is the patient set which includes all patients who were documented to have taken at least one dose of treatment and who had a baseline HbA1c value at at least one on-treatment HbA1c.
Measure: Mean (Standard Error); unit: percent
Groups:
- Pio15: Participants treated with pioglitazone 15mg monotherapy for the first 30 weeks
- Pio30: Participants treated with pioglitazone 30mg monotherapy for the first 30 weeks
- Pio45: Participants treated with pioglitazone 30mg monotherapy for 6 weeks and were titrated to pioglitazone 45mg monotherapy for the next 24 weeks.
- Lina5: Participants treated with linagliptin 5mg once daily for the first 30 weeks
- Lina5Pio15: Participants treated with linagliptin 5mg + pioglitazone 15mg fixed dose combination (FDC) for the first 30 weeks
- Lina5Pio30: Participants treated with linagliptin 5mg + pioglitazone 30mg fixed dose combination (FDC) for the first 30 weeks
- Lina5Pio45: Participants treated with linagliptin 5mg + pioglitazone 30mg fixed dose combination (FDC) for the first 6 weeks and were titrated to linagliptin 5mg + pioglitazone 45mg for the next 24 weeks.
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 124 | 134 | 134 | 130 | 120 | 125 | 126
percent | -0.66 (0.09) | -0.69 (0.09) | -0.87 (0.09) | -0.39 (0.09) | -0.83 (0.09) | -1.06 (0.09) | -1.28 (0.09)
Statistical Analysis 1: Comparison: Pio15 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.1571, ANCOVA — The model includes fixed effects for treatment, continuous baseline HbA1c, prior anti-diabetic medication and country; Mean Difference (Final Values) = -0.17, 95% CI [-0.41 to 0.07]
Statistical Analysis 2: Comparison: Pio30 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0016, ANCOVA; The model includes fixed effects for treatment, continuous baseline HbA1c, prior anti-diabetic medication and country; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.60 to -0.14]
Statistical Analysis 3: Comparison: Pio45 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0006, ANCOVA; The model includes fixed effects for treatment, continuous baseline HbA1c, prior anti-diabetic medication and country; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.64 to -0.18]
Statistical Analysis 4: Comparison: Lina5 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0003, ANCOVA; The model includes fixed effects for treatment, continuous baseline HbA1c, prior anti-diabetic medication and country; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.67 to -0.20]
Statistical Analysis 5: Comparison: Lina5 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; The model includes fixed effects for treatment, continuous baseline HbA1c, prior anti-diabetic medication and country; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-0.91 to -0.44]
Statistical Analysis 6: Comparison: Lina5 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; The model includes fixed effects for treatment, continuous baseline HbA1c, prior anti-diabetic medication and country; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-1.12 to -0.66]

2. Secondary Outcome: Occurrence of Cumulative Treat to Target Efficacy Response, of HbA1c Under Treatment of < 7.0% After 30 Weeks of Treatment
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin.
Time Frame: Baseline and 30 weeks
Population: FAS patients who also had baseline HbA1c>=7%.Non-completers (patients without a value at Week 30) were considered as failures (NCF).
Measure: Number; unit: participants
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 121 | 125 | 129 | 124 | 112 | 118 | 121
participants | 39 | 55 | 68 | 29 | 45 | 61 | 81
Statistical Analysis 1: Comparison: Pio15 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.4639, Regression, Logistic; A logistic regression model with terms for treatment, continuous HbA1c baseline, prior use of antidiabetic agents and country; Odds Ratio (OR) = 1.246, 95% CI [0.692 to 2.242]
Statistical Analysis 2: Comparison: Pio30 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0546, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.746, 95% CI [0.989 to 3.083]
Statistical Analysis 3: Comparison: Pio45 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0254, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.903, 95% CI [1.083 to 3.345]
Statistical Analysis 4: Comparison: Lina5 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0009, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.804, 95% CI [1.524 to 5.159]
Statistical Analysis 5: Comparison: Lina5 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 5.429, 95% CI [2.947 to 10.001]
Statistical Analysis 6: Comparison: Lina5 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 9.614, 95% CI [5.187 to 17.821]

3. Secondary Outcome: Occurrence of Cumulative Treat to Target Efficacy Response, of HbA1c Under Treatment of < 6.5% After 30 Weeks of Treatment
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin.
Time Frame: Baseline and 30 weeks
Population: FAS patients who also had baseline HbA1c >=6.5%. Non-completers (patients without a value at Week 30) were considered as failures (NCF)
Measure: Number; unit: participants
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 124 | 132 | 134 | 129 | 120 | 123 | 125
participants | 20 | 28 | 39 | 14 | 24 | 38 | 43
Statistical Analysis 1: Comparison: Pio15 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.7359, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.126, 95% CI [0.565 to 2.243]
Statistical Analysis 2: Comparison: Pio30 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0363, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.905, 95% CI [1.042 to 3.484]
Statistical Analysis 3: Comparison: Pio45 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.4039, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.269, 95% CI [0.726 to 2.217]
Statistical Analysis 4: Comparison: Lina5 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0345, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.220, 95% CI [1.060 to 4.649]
Statistical Analysis 5: Comparison: Lina5 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 4.580, 95% CI [2.263 to 9.266]
Statistical Analysis 6: Comparison: Lina5 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 5.066, 95% CI [2.530 to 10.145]

4. Secondary Outcome: Occurrence of Relative Efficacy Response (HbA1c Lowering by at Least 0.5% After 30 Weeks of Treatment)
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin.
Time Frame: Baseline and 30 weeks
Population: FAS with non-completers (without a value at Week 30) considered as failure
Measure: Number; unit: participants
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 124 | 134 | 134 | 130 | 120 | 125 | 126
participants | 79 | 83 | 90 | 54 | 79 | 91 | 107
Statistical Analysis 1: Comparison: Pio15 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.7540, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.090, 95% CI [0.637 to 1.863]
Statistical Analysis 2: Comparison: Pio30 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0506, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.707, 95% CI [0.999 to 2.918]
Statistical Analysis 3: Comparison: Pio45 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.966, 95% CI 2-sided [1.604 to 5.485]
Statistical Analysis 4: Comparison: Lina5 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.696, 95% CI [1.594 to 4.559]
Statistical Analysis 5: Comparison: Lina5 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 4.017, 95% CI [2.348 to 6.873]
Statistical Analysis 6: Comparison: Lina5 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 8.521, 95% CI [4.630 to 15.681]

5. Secondary Outcome: HbA1c Change From Baseline by Visit Over Time
Description: HbA1c is measured as a percentage. The change from baseline is the HbA1c over time minus the baseline HbA1c. The model includes fixed effects for treatment, continuous baseline HbA1c, prior andi-diabetic medication, country, visit and treatment.
  by visit interaction.
Time Frame: Baseline, week 6, week 12, week 18, week 24, week 30
Population: FAS (observed cases)
Measure: Mean (Standard Error); unit: percent
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 124 | 134 | 134 | 130 | 120 | 125 | 126
percent
  Change to week 6 (N=121,133,133,130,119,124,125) | -0.22 (0.06) | -0.16 (0.06) | -0.20 (0.06) | -0.23 (0.06) | -0.43 (0.06) | -0.47 (0.06) | -0.62 (0.06)
  Change to week 12 (N=112,124,127,122,111,117,120) | -0.47 (0.08) | -0.43 (0.07) | -0.59 (0.07) | -0.36 (0.08) | -0.71 (0.08) | -0.92 (0.08) | -1.01 (0.08)
  Change to week 18 (N=101,121,122,112,104,104,115) | -0.63 (0.09) | -0.58 (0.08) | -0.82 (0.08) | -0.39 (0.08) | -0.81 (0.09) | -1.07 (0.09) | -1.22 (0.09)
  Change to week 24 (N=91,108,110,95,92,96,109) | -0.75 (0.09) | -0.67 (0.09) | -0.87 (0.09) | -0.39 (0.09) | -0.84 (0.09) | -1.10 (0.09) | -1.23 (0.09)
  Change to week 30 (N=78,93,91,79,86,87,97) | -0.77 (0.09) | -0.73 (0.08) | -0.94 (0.09) | -0.37 (0.09) | -0.87 (0.09) | -1.09 (0.09) | -1.27 (0.09)

6. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline After 30 Weeks of Treatment
Description: The change from baseline is the FPG after 30 weeks minus the baseline FPG.
Time Frame: Baseline and 30 weeks
Population: Patients from Full Analysis Set (FAS) with a value for FPG at baseline and on-treatment. Last observation carried forward (LOCF) used to handle missing values at Week 30.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 123 | 133 | 134 | 130 | 119 | 123 | 125
mg/dL | -15.16 (3.49) | -25.49 (3.28) | -28.69 (3.29) | -1.46 (3.35) | -18.84 (3.47) | -27.33 (3.46) | -35.19 (3.40)
Statistical Analysis 1: Comparison: Pio15 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.4275, ANCOVA; The model includes fixed effects for treatment, continuous baseline HbA1c, continuous baseline FPG, prior anti-diabetic medication and country; Mean Difference (Final Values) = -3.68, 95% CI 2-sided [-12.77 to 5.42]
Statistical Analysis 2: Comparison: Pio30 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.6839, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.84, 95% CI 2-sided [-10.69 to 7.02]
Statistical Analysis 3: Comparison: Pio45 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.1466, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -6.50, 95% CI 2-sided [-15.29 to 2.28]
Statistical Analysis 4: Comparison: Lina5 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0002, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -17.38, 95% CI 2-sided [-26.35 to -8.41]
Statistical Analysis 5: Comparison: Lina5 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -25.87, 95% CI 2-sided [-34.77 to -16.98]
Statistical Analysis 6: Comparison: Lina5 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -33.73, 95% CI 2-sided [-42.57 to -24.89]

7. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline by Visit Over Time
Description: The change from baseline is the FPG over time minus the baseline FPG. Model includes fixed effects for treatment, continuous baseline FPG, continuous baseline HbA1c, prior anti-diabetic medication, country, visit and treatment by visit interaction
Time Frame: Baseline, week 6, week 12, week 18, week 24, week 30
Population: FAS (observed cases)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 124 | 134 | 134 | 130 | 120 | 125 | 126
mg/dL
  Change at week 6 (N=118,132,133,130,119,122,124) | -14.43 (2.99) | -16.38 (2.80) | -15.72 (2.81) | -4.25 (2.84) | -19.25 (2.96) | -26.89 (2.94) | -28.36 (2.89)
  Change at week 12 (N=111,124,126,122,108,114,118) | -10.63 (3.24) | -21.36 (3.04) | -25.30 (3.03) | -7.43 (3.08) | -17.99 (3.24) | -31.25 (3.19) | -28.53 (3.13)
  Change at week 18 (N=100,122,121,111,104,103,114) | -16.68 (3.29) | -20.69 (3.02) | -28.68 (3.03) | -7.06 (3.13) | -19.01 (3.24) | -31.22 (3.25) | -30.66 (3.12)
  Change at week 24 (N=90,108,108,96,93,93,108) | -16.25 (3.25) | -21.57 (2.99) | -27.67 (3.00) | -4.60 (3.13) | -16.68 (3.20) | -31.48 (3.20) | -31.49 (3.03)
  Change at week 30 (N=76,91,89,79,82,87,98) | -17.66 (3.35) | -26.09 (3.08) | -31.76 (3.11) | -0.09 (3.24) | -17.93 (3.27) | -27.11 (3.22) | -34.04 (3.07)

8. Secondary Outcome: Two-hour Postprandial Glucose (2hPPG) Change From Baseline at Week 30 by Meal Tolerance Test (MTT)
Description: The change from baseline is the 2hPPG after 30 weeks minus the baseline 2hPPG.
Time Frame: Baseline and 30 weeks
Population: MTT set: This patient set includes those patients in the FAS who had a valid MTT at baseline and at least one valid on-treatment MTT. An MTT is considered valid if both an FPG and a 2-hour PPG value are available.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 29 | 34 | 25 | 22 | 28 | 26 | 31
mg/dL | -30.65 (10.93) | -83.00 (9.85) | -82.98 (10.92) | -51.61 (11.67) | -67.26 (11.15) | -87.94 (11.14) | -84.77 (10.28)
Statistical Analysis 1: Comparison: Pio15 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0057, ANCOVA; The model includes fixed effects for treatment, continuous baseline HbA1c and 2-hour PPG, prior anti-diabetic medication and country; Mean Difference (Final Values) = -36.61, 95% CI 2-sided [-62.42 to -10.80]
Statistical Analysis 2: Comparison: Pio30 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.7021, ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -4.94, 95% CI [-30.39 to 20.51]
Statistical Analysis 3: Comparison: Pio45 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.8932, ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.78, 95% CI 2-sided [-27.95 to 24.38]
Statistical Analysis 4: Comparison: Lina5 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.2706, ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -15.65, 95% CI 2-sided [-43.60 to 12.30]
Statistical Analysis 5: Comparison: Lina5 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0126, ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -36.33, 95% CI 2-sided [-64.78 to -7.89]
Statistical Analysis 6: Comparison: Lina5 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0167, ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -33.16, 95% CI 2-sided [-60.23 to -6.08]

9. Secondary Outcome: Time to First Use of Rescue Therapy
Description: Proportion of patients at 30 weeks with rescue therapy using Kaplan-Meier analysis.
Time Frame: 30 weeks
Population: FAS
Measure: Number; unit: Proportion of participants
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 124 | 134 | 134 | 130 | 120 | 125 | 126
Proportion of participants
  Proportion event-free | 0.8117 (50.5) | 0.8533 (47.8) | 0.9051 (55.3) | 0.7756 (47.7) | 0.8854 (61.5) | 0.9078 (54.7) | 0.9548 (65.7)
  Standard Error | 0.0382 | 0.0330 | 0.0273 | 0.0390 | 0.0313 | 0.0279 | 0.0198

10. Secondary Outcome: Incidence of Rescue Therapy During the First 30 Weeks of Treatment
Description: Rescue therapy was defined to include any new antidiabetic medication taken for hyperglycemia and introduced on or after the start date of study treatment and before the end date of study treatment.
Time Frame: 30 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Pio15 | Pio30 | Pio45 | Lina5 | Lina5Pio15 | Lina5Pio30 | Lina5Pio45
Number analyzed (Participants) | 124 | 134 | 134 | 130 | 120 | 125 | 126
participants | 20 | 17 | 11 | 26 | 12 | 10 | 5
Statistical Analysis 1: Comparison: Pio15 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.3052, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.649, 95% CI [0.284 to 1.482]
Statistical Analysis 2: Comparison: Pio30 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0844, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.456, 95% CI 2-sided [0.187 to 1.112]
Statistical Analysis 3: Comparison: Pio45 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.1561, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.443, 95% CI 2-sided [0.143 to 1.365]
Statistical Analysis 4: Comparison: Lina5 vs Lina5Pio15; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0146, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.368, 95% CI [0.165 to 0.821]
Statistical Analysis 5: Comparison: Lina5 vs Lina5Pio30; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0009, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.238, 95% CI [0.102 to 0.557]
Statistical Analysis 6: Comparison: Lina5 vs Lina5Pio45; Treatment comparisons are for fixed dose combination versus monotherapy; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.141, 95% CI [0.050 to 0.397]

ADVERSE EVENTS:
Time Frame: Up to 85 weeks
Arm/Group | Pio15/Pio30 | Pio30/Pio30 | Pio45/Pio45 | Lina5/Lina5 | Lina5Pio15/Lina5Pio30 | Lina5Pio30/Lina5Pio30 | Lina5Pio45/Lina5Pio45
Serious Adverse Events (participants affected / at risk) | 9/131 | 9/140 | 5/138 | 9/135 | 9/126 | 15/133 | 10/133
Other Adverse Events (participants affected / at risk) | 57/131 | 55/140 | 66/138 | 57/135 | 52/126 | 58/133 | 56/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pio15/Pio30 (N=131) | Pio30/Pio30 (N=140) | Pio45/Pio45 (N=138) | Lina5/Lina5 (N=135) | Lina5Pio15/Lina5Pio30 (N=126) | Lina5Pio30/Lina5Pio30 (N=133) | Lina5Pio45/Lina5Pio45 (N=133)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal artery embolism (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Encephalitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric bypass (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vascular graft (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pio15/Pio30 (N=131) | Pio30/Pio30 (N=140) | Pio45/Pio45 (N=138) | Lina5/Lina5 (N=135) | Lina5Pio15/Lina5Pio30 (N=126) | Lina5Pio30/Lina5Pio30 (N=133) | Lina5Pio45/Lina5Pio45 (N=133)
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 5 | 7 | 10 | 2 | 3
Oedema (General disorders) | 4 | 1 | 7 | 0 | 0 | 12 | 4
Oedema peripheral (General disorders) | 13 | 11 | 11 | 6 | 8 | 9 | 15
Bronchitis (Infections and infestations) | 5 | 4 | 7 | 4 | 3 | 2 | 5
Nasopharyngitis (Infections and infestations) | 9 | 10 | 4 | 10 | 9 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 9 | 5 | 4 | 6 | 6
Urinary tract infection (Infections and infestations) | 7 | 7 | 8 | 8 | 5 | 7 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 10 | 5 | 14 | 8 | 8 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 9 | 7 | 1 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 5 | 10 | 6 | 8 | 7 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 5 | 3 | 7 | 7 | 6
Dizziness (Nervous system disorders) | 0 | 7 | 3 | 4 | 4 | 9 | 4
Headache (Nervous system disorders) | 7 | 7 | 9 | 6 | 5 | 5 | 6
Hypertension (Vascular disorders) | 12 | 4 | 7 | 9 | 6 | 5 | 1

LIMITATIONS AND CAVEATS:
The study (Part B treatment only) was stopped early by protocol amendment #5, although Part A (time frame for all efficacy outcomes) proceeded to completion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.